CLINICAL TRIAL: NCT07355491
Title: Performance Evaluation of Dream OCT: AP Study
Status: Recruiting | Type: Observational
Sponsor: Intalight, Inc (Industry)
Collaborators: Illinois College of Optometry (Other)
Responsible Party: Sponsor
Other Study IDs: DREAM-CP2025-001
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Glaucoma Patients; Retina Patients; Eyes With Corneal Abnormality; Normal Healthy Eyes
Keywords: Eyes with ocular pathology and normal healthy eyes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Normal Healthy Eyes: Eyes without pathology
  Interventions: Device: This is an observational study only, all patients are imaged on the investigational device
- Glaucoma: Patients with glaucoma in one or both eyes
  Interventions: Device: This is an observational study only, all patients are imaged on the investigational device
- Retina: Patients with retina pathology in one or both eyes
  Interventions: Device: This is an observational study only, all patients are imaged on the investigational device
- Cornea: Eyes with cornea abnormality in one or both eyes
  Interventions: Device: This is an observational study only, all patients are imaged on the investigational device

INTERVENTIONS:
Device: This is an observational study only, all patients are imaged on the investigational device — This study is a non-significant risk study where enrolled patients are imaged on an investigational device and a predicate device

SUMMARY:
This study will evaluate the clinical performance of a new swept-source OCT imaging device, the VG200D, and to evaluate substantial equivalence with a predicate device, the Cirrus 5000. Clinical performance will be assessed through an agreement and precision analysis of OCT measurement parameters.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the clinical performance of a new swept-source OCT imaging device, the VG200D, and to evaluate substantial equivalence with a predicate device, the Cirrus 5000. Clinical performance will be assessed through an agreement and precision analysis of OCT measurement parameters. Evidence for substantial equivalence will be through establishing equivalent precision results between devices and meeting pre-determined performance goals for precision and agreement results for a majority of parameters.

The primary objective of this study is to evaluate agreement and precision of measurements between the VG200D and the predicate device Cirrus.

Primary endpoints include the agreement and precision results from the Anterior Segment OCT measurements for cornea and epithelial thickness in normal eyes and eyes with a corneal abnormality and the posterior segment OCT measurements for the retina, ganglion cell +IPL, RNFL, and optic nerve in normal eyes, eyes with glaucoma, and eyes with retinal pathology.

This is a prospective comparative study that will be conducted at one clinical site in the United States, in which subjects who sign an informed consent form and fulfil all inclusion and exclusion criteria will have images obtained using the study device and the predicate device (VG200D and Cirrus respectively).

Subjects enrolled in this study will be confirmed to have normal healthy eyes, eyes with retina pathology, eyes with glaucoma, or eyes with cornea abnormality. Ocular status will be determined by a thorough clinical examination after enrollment. Except for normal eyes, subjects enrolled may have more than one ocular pathology. If subjects have more than one ocular pathology, the investigator will enroll them in the study group based on the ocular pathology that is more clinically significant (more severe).

There will be two main types of analyses performed as part of this study, including 1) a precision analysis, and 2) an agreement analysis.

ELIGIBILITY:
Inclusion Criteria for Normal Group:

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects with normal eye examinations in both eyes on the date of the study visit as observed with a 90 diopter lens
4. BCVA 20/40 or better (each eye) on the date of the study visit

Exclusion Criteria for Normal Group:

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects not able to obtain acceptable OCT images due to ocular media opacity or other reasons
3. Subject has a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
4. Presence of any ocular pathology except for cataract in either eye

Inclusion Criteria for Glaucoma Group:

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. BCVA 20/40 or better in the study eye
4. History of Visual field defects within the previous year from the study visit or measured the day of the study visit consistent with glaucomatous optic nerve damage with at least one of the following two findings:

   1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
   2. Glaucoma hemi-field test "outside normal limits."
5. Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities:

   1. Diffuse thinning, focal narrowing, or notching of the neuroretinal rim, especially at the inferior or superior poles with or without disc hemorrhage;
   2. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue

Exclusion Criteria for Glaucoma Group:

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects not able to obtain acceptable OCT images due to ocular media opacity or other reasons
3. Subject has a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
4. No reliable Humphrey Field Analyzer (HFA) visual field (24-2 SITA Standard or Fast, 10-2, white on white) result within the past year of the study visit, defined as fixation losses > 33%, or false positives > 33%, or false negatives > 33% in the study eye

Inclusion Criteria for Retina Disease Group:

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. BCVA 20/400 or better in the study eye
4. Diagnosis of some type of retinal pathology by investigator, may include, but not limited to: Macular Degeneration (including patients with drusen and geographic atrophy and choroidal neovascularization), Diabetic Macular Edema, Diabetic Retinopathy, Macular Hole, Epiretinal Membrane, Central Serous Retinopathy, Vein or artery Occlusions and others

Exclusion Criteria for Retinal Disease Group:

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects not able to obtain acceptable OCT images due to ocular media opacity or other reasons
3. Subject has a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Inclusion Criteria for Cornea Group:

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects with one of the following corneal abnormalities:

   i. Cornea disease (e.g., Fuch's or other) ii. Keratoconus iii. Cornea transplant iv. Post refractive surgery (e.g., LASIK or other) v. Dry Eye Syndrome vi. Long-term contact wearers (greater than 1 year)
4. BCVA 20/400 or better in the study eye

Exclusion Criteria for Cornea Group:

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects not able to obtain acceptable OCT images due to ocular media opacity or other reasons
3. Subject has a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population includes patients with normal healthy eyes, patients with glaucoma, patients with retina pathology and patients with abnormal corneas
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Agreement results and Precision Results | This study will last approximately 6 months
  Primary endpoints include the agreement and precision results from the Anterior Segment OCT measurements for cornea and epithelial thickness in normal eyes and eyes with a corneal abnormality and the posterior segment OCT measurements for the retina, ganglion cell +IPL, RNFL, and optic nerve in normal eyes, eyes with glaucoma, and eyes with retinal pathology.

SECONDARY OUTCOMES:
Device Safety | the study duration is approximately 6 months
  Any and all adverse events associated with this study will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Micahel Chaglasian, OD, Principal Investigator — Illinois College of Optometry
Locations (1):
- Illinois College of Optometry, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The study data will be used for an FDA 510k filing